CLINICAL TRIAL: NCT03366337
Title: A Phase 2 Trial of the Safety and Efficacy of Bardoxolone Methyl in Patients With Rare Chronic Kidney Diseases
Brief Title: A Phase 2 Trial of the Safety and Efficacy of Bardoxolone Methyl in Patients With Rare Chronic Kidney Diseases - PHOENIX
Acronym: PHOENIX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1702
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: IgA Nephropathy; CKD Associated With Type 1 Diabetes; Focal Segmental Glomerulosclerosis; Autosomal Dominant Polycystic Kidney
Keywords: IgA Nephropathy; CKD associated with type 1 diabetes; Focal segmental glomerulosclerosis; Autosomal dominant polycystic kidney disease; IgAN; FSGS; ADPKD; Bardoxolone methyl; CDDO-ME; RTA 402
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental; Polycystic Kidney, Autosomal Dominant | interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bardoxolone Methyl - ADPKD (Experimental): Participants with autosomal polycystic kidney disease (ADPKD) will receive bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Interventions: Drug: Bardoxolone methyl capsules
- Bardoxolone Methyl - IgAN (Experimental): Participants with IgA nephropathy (IgAN) will receive bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Interventions: Drug: Bardoxolone methyl capsules
- Bardoxolone Methyl - T1D (Experimental): Participants with Type 1 diabetes (T1D) will receive bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Interventions: Drug: Bardoxolone methyl capsules
- Bardoxolone Methyl - FSGS (Experimental): Participants with focal segmental glomerulosclerosis (FSGS) will receive bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Interventions: Drug: Bardoxolone methyl capsules

INTERVENTIONS:
Drug: Bardoxolone methyl capsules — Bardoxolone 5 mg capsules
  Other Names: RTA 402

SUMMARY:
This multi-center, open-label Phase 2 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with the following rare chronic kidney diseases (CKD): CKD associated with type 1 diabetes (T1D), IgA nephropathy (IgAN), focal segmental glomerulosclerosis (FSGS), and autosomal dominant polycystic kidney disease (ADPKD). Patients will be enrolled in disease specific cohorts within the trial, and effectiveness of bardoxolone methyl in treating CKD will be assessed separately by cohort for each rare CKD.

All patients in the study will follow the same visit and assessment schedule. Following randomization on Day 1, patients will be scheduled to be assessed during treatment at Weeks 1, 2, 4, 6, 8, and 12, and by telephone contact on Days 3, 10, 21, 31, 38, and 45. Patients will also be scheduled to be assessed at an in-person follow-up visit at Week 16, four weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 ≤ age ≤ 65 upon study consent;
* Screening eGFR (average of Screen A and Screen B eGFR values) ≥ 30 and ≤ 90 mL/min/1.73 m2. The two eGFR values collected at Screen A and Screen B visits used to determine eligibility must have a percent difference ≤ 25%;
* Albumin to creatinine ratio (ACR) ≤ 2500 mg/g at Screen B visit;
* If receiving an angiotensin-converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB), patients should be prescribed the maximally tolerated labeled daily dose (MTLDD) for at least 6 weeks prior to the Screen A visit;
* For patients enrolling in T1D Cohort: Diagnosis of type 1 diabetes confirmed by fasting C-peptide level. Diagnosis must have been made ≤ 35 years of age; and prescribed stable dose of insulin to maintain adequate glucose control for at least 6 months prior to the Screen A visit;
* For patients enrolling in IgAN Cohort: Biopsy-confirmed IgA nephropathy;
* For patients enrolling in FSGS Cohort: Biopsy-confirmed FSGS that is not due to known secondary causes including morbid obesity, decreased renal mass, viral infections, drug-induced nephrotoxicity, or prior history of vasculitis;
* For patients enrolling in ADPKD Cohort: Genetic confirmation of PKD1 mutation;
* Adequate bone marrow reserve and organ function at the Screen A visit as follows: Hematologic: Absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L, hemoglobin (Hgb) ≥ 9 g/dL; and Hepatic: Total bilirubin (TBL) ≤ 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times ULN.

Exclusion Criteria:

* Kidney or any other solid organ transplant recipient or a planned transplant during the study;
* B-type natriuretic peptide (BNP) level > 200 pg/mL at Screen A visit;
* Acute dialysis or acute kidney injury within 12 weeks prior to Screen A visit or during Screening;
* Serum albumin < 3 g/dL at Screen A visit;
* Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to randomization or anticipated need for immunosuppression during the study;
* For patients enrolling in IgAN Cohort: Systemic manifestations of Henoch-Schonlein purpura within 1 year prior to Screen A visit; or have used belimumab, eculizumab, or rituximab within 6 months prior to Screen A visit;
* For patients enrolling in ADPKD Cohort: Receiving tolvaptan;
* Cerebrovascular event (stroke, transient ischemic attack) or aneurysm within 6 months prior to Screen A visit or during Screening;
* History of clinically significant left-sided heart disease and/or clinically significant cardiac disease;
* Uncontrolled systemic hypertension;
* Systolic BP < 90 mm Hg at Screen A visit after a period of rest;
* History of malignancy within 2 years prior to Screen A visit, with the exception of localized skin or cervical carcinomas;
* Uncontrolled diabetes (HbA1c > 10.0%) at Screen A visit;
* Untreated or uncontrolled active bacterial, fungal, or viral infection;
* Participation in other interventional clinical studies within 30 days prior to Day 1;
* Unwilling to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential) during Screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested;
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Phoenician Centers for Research & Innovation (PCRI), Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Denver Nephrology, Denver, Colorado
  - Gulfcoast Endocrine and Diabetes Center, Clearwater, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Coastal Nephrology Associates, Port Charlotte, Florida
  - Kidney Care Augusta, Augusta, Georgia
  - Boise Kidney & Hypertension, PLLC, Caldwell, Idaho
  - Boise Kidney & Hypertension, PLLC, Meridian, Idaho
  - Research By Design, Evergreen Park, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Tufts Medical Center - Division of Nephrology Tufts Medical Center, Boston, Massachusetts
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center - Nephrology, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Physician's East Endocrine Research, Greenville, North Carolina
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - The Warren Alpert School of Brown University, Providence, Rhode Island
  - Nephrology Associates, Chattanooga, Tennessee
  - Research Management, Inc., Austin, Texas
  - Renal Disease Research Intitute, Dallas, Texas
  - Renal Associates, PA, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Mendez Center for Clinical Research LLC, Fairfax Station, Virginia
  - Larry Stonesifer, M.D., Federal Way, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bardoxolone Methyl - ADPKD: Participants with autosomal polycystic kidney disease (ADPKD) who received bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Bardoxolone methyl capsules: Bardoxolone 5 mg capsules
- Bardoxolone Methyl - IgAN: Participants with IgA nephropathy (IgAN) who received bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Bardoxolone methyl capsules: Bardoxolone 5 mg capsules
- Bardoxolone Methyl - T1D: Participants with Type 1 diabetes (T1D) who received bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Bardoxolone methyl capsules: Bardoxolone 5 mg capsules
- Bardoxolone Methyl - FSGS: Participants with focal segmental glomerulosclerosis (FSGS) who received bardoxolone methyl capsules at a starting dose of 5 mg and titrate up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily.
  Bardoxolone methyl capsules: Bardoxolone 5 mg capsules
Period: Overall Study
Arm/Group | Bardoxolone Methyl - ADPKD | Bardoxolone Methyl - IgAN | Bardoxolone Methyl - T1D | Bardoxolone Methyl - FSGS
Started | 31 | 26 | 28 | 18
Completed | 28 | 26 | 26 | 17
Not Completed | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received any amount of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Bardoxolone Methyl - ADPKD | Bardoxolone Methyl - IgAN | Bardoxolone Methyl - T1D | Bardoxolone Methyl - FSGS | Total
Number analyzed (Participants) | 31 | 26 | 28 | 18 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.49) | 48.5 (9.53) | 49 (9.91) | 48.6 (12.79) | 48.3 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 11 | 21 | 10 | 63
  Male | 10 | 15 | 7 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 1 | 8
  Not Hispanic or Latino | 28 | 24 | 26 | 17 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 4 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 5 | 10
  White | 25 | 22 | 27 | 11 | 85
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — eGFR is a measure of kidney function assessed through blood/serum. Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function.
  mL/min/1.73 m^2 | 47.69 (13.630) | 46.19 (12.576) | 67.52 (17.059) | 51.66 (18.144) | 53.39 (17.427)
Baseline urine albumin-to-creatinine ratio (UACR) [Mean (Full Range); unit: mg/g] — UACR (urine albumin-to-creatinine ratio) is a marker of kidney health, and an increase in UACR is observed with kidney diseases of multiple etiologies. Lower UACR values represent improved kidney function.
  mg/g | 44.40 [2.4 to 1824.5] | 104.03 [5.2 to 1288.0] | 30.88 [2.5 to 1208.0] | 184.30 [3.5 to 1006.5] | 63.95 [2.4 to 1824.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 12
Description: To assess the change in eGFR from baseline to week 12. eGFR is a measure of kidney function assessed through blood/serum. Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function.
Time Frame: 12 weeks after participant receives the first dose
Population: Intent-to-treat population (all enrolled patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Bardoxolone Methyl - ADPKD | Bardoxolone Methyl - IgAN | Bardoxolone Methyl - T1D | Bardoxolone Methyl - FSGS
Number analyzed (Participants) | 31 | 26 | 28 | 18
mL/min/1.73 m^2 | 9.31 (1.3743) | 8.00 (1.5700) | 5.46 (2.2792) | 7.83 (2.216)
Statistical Analysis 1: Comparison: Bardoxolone Methyl - ADPKD; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 12; p < 0.0001, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 12 were included. Missing data were not imputed; LS Mean change from baseline = 9.31, 95% CI 2-sided [6.5 to 12.13], Standard Error of Mean 1.3743
Statistical Analysis 2: Comparison: Bardoxolone Methyl - IgAN; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 12; p < 0.0001, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 12 were included. Missing data were not imputed; LS Mean change from baseline = 8.00, 95% CI 2-sided [4.75 to 11.25], Standard Error of Mean 1.5700
Statistical Analysis 3: Comparison: Bardoxolone Methyl - T1D; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 12; p = 0.0247, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 12 were included. Missing data were not imputed; LS Mean change from baseline = 5.46, 95% CI 2-sided [0.76 to 10.16], Standard Error of Mean 2.2792
Statistical Analysis 4: Comparison: Bardoxolone Methyl - FSGS; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 12; p = 0.0030, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 12 were included. Missing data were not imputed; LS Mean change from baseline = 7.83, 95% CI 2-sided [3.11 to 12.55], Standard Error of Mean 2.2160

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: After the first dose, documentation of adverse events was to continue until 30 days (+/- 3 days) following administration of the final dose of study medication, regardless of the relationship of the adverse event to study drug.
Arm/Group | Bardoxolone Methyl - ADPKD | Bardoxolone Methyl - IgAN | Bardoxolone Methyl - T1D | Bardoxolone Methyl - FSGS
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/26 | 0/28 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/26 | 0/28 | 1/18
Other Adverse Events (participants affected / at risk) | 30/31 | 22/26 | 25/28 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl - ADPKD (N=31) | Bardoxolone Methyl - IgAN (N=26) | Bardoxolone Methyl - T1D (N=28) | Bardoxolone Methyl - FSGS (N=18)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl - ADPKD (N=31) | Bardoxolone Methyl - IgAN (N=26) | Bardoxolone Methyl - T1D (N=28) | Bardoxolone Methyl - FSGS (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 5 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 5 | 4 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 3 | 2
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Adenoviral upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 1 | 2 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 3 | 3 | 2
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 2 | 0 | 0 | 0
Transaminases increased (Investigations) | 2 | 4 | 2 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 9 | 9 | 9
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Aura (Nervous system disorders) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 5 | 6 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03366337/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT03366337/SAP_001.pdf